CLINICAL TRIAL: NCT05230927
Title: Cognitive Impairment, Frailty and Rehabilitative Outcome in Older Patients Affected by Cardiorespiratory Disease (DEC_FRAinRIAB)
Brief Title: Cognitive Impairment, Frailty and Rehabilitative Outcome in Older Patients Affected by Cardiorespiratory Disease
Status: Completed | Type: Observational
Sponsor: Antonia Pierobon (Other)
Responsible Party: Sponsor-Investigator, Antonia Pierobon, Principal investigator, Istituti Clinici Scientifici Maugeri SpA
Organization: Istituti Clinici Scientifici Maugeri SpA (Other)
Other Study IDs: 2424
Record Dates: First submitted 2021-12-31; First posted 2022-02-09 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Chronic Heart Failure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Heart Failure
  Interventions: Other: Multidisciplinary Rehabilitation
- Chronic Obstructive Pulmonary Disease
  Interventions: Other: Multidisciplinary Rehabilitation

INTERVENTIONS:
Other: Multidisciplinary Rehabilitation — All patients admitted to an inpatient rehabilitation program will undergo medical history collection, physical, clinical, and functional examination, exercise testing, educational sessions, exercise training (cycle ergometer/treadmill, arm ergometer, breathing, and strength exercises where indicated, calisthenics exercises), psychological counseling, and metabolic evaluation with a personalized diet when needed.

SUMMARY:
A consistent number of studies in the last few years highlighted that the functional and clinical worsening in patients with cardiac and/or respiratory disease/s increase the risk of cognitive decline.

The literature reports a greater diffusion of screening procedures for cognitive deficits in patients with cardiac diseases compared to patients with respiratory diseases. However, in both populations, the interest for cognitive impairment is justified by multiple reasons: the numerous exacerbations of the disease and re-hospitalizations, the difficulty in following complex therapeutic regimens and recognizing worsening of symptoms, the reduced functional autonomy and the rehabilitation outcome . Although recently the Italian Society of Geriatrics and Gerontology has raised the threshold for the definition of the 'elderly' patient from 65 to 75 years to better adapt to the current physical and mental performance of men and women living in economically developed countries and to the demographic situation of the Italian population. Therefore the three classes of 'elderly' patients that we will enroll will be defined as follows: "young old" (65-74 years), "old" (75-84 years), and "old-old" (≥85 years). In general, the age of the eligible sample is defined as ≥ 65 years.

Furthermore, in chronic diseases, emotional factors, such as anxiety and depression, also play an important role in disease adaptation and in the rehabilitation outcome in both cardiac and respiratory diseases.

Alongside the problems relating to emotional aspects and cognitive decline, the frailty syndrome is noteworthy, particularly in the elderly and in the presence of cardiac/respiratory diseases. Frailty is associated with the loss of functionality that leads to greater vulnerability to adverse events such as the increased risk of falls, hospitalization, institutionalization, disability and mortality.

Frailty screening or assessment scales provide predictive information on the risk of death and institutionalization and they are a good predictor of acute hospital outcomes too. Instead, concerning what emerges from international literature, in rehabilitation cardiology, despite the increase in the presence of elderly patients, the clinical and prognostic relevance of frailty has not yet been well defined and measured. On the other hand, recent studies points out that frailty is present in 1/4 of outpatient COPD patients, it is an independent predictor of rehabilitation program interruption and it is also easily reversible in the short term after rehabilitation, thus frailty appears to be one of the relevant aspects in rehabilitative treatment.

In light of the data in the literature, the purposes of this prospective observational study are to evaluate the following objectives:

1. At baseline, the presence of cognitive impairment, anxiety, depression, the assessment of self-reported adherence to therapeutic prescriptions and frailty in a sample of elderly patients (age ≥65) with chronic cardiorespiratory disease admitted for a cardiorespiratory rehabilitation cycle and the correlation with disease severity and functional aspects.
2. In follow-up, the impact that these factors have on the rehabilitation outcome at the end of hospitalization and on the state of health at six months (telephone interview).

ELIGIBILITY:
Inclusion Criteria:

All inpatients admitted to the Cardiac Rehabilitation Department and the Pulmonary Rehabilitation Department of ICS Maugeri - Tradate (Varese) and Montescano (Pavia) affected by CHF or COPD.

Exclusion Criteria:

* severe clinical conditions (chronic inflammatory diseases, neoplasia)
* psychiatric and neurological conditions(at anamnestic or actual clinical evaluation),
* no Italian education, illiteracy or relapse into illiteracy,
* severe visuo-perceptive deficits,
* lack of motivation or refusal to undergo the evaluation,
* severe cognitive deterioration (Mini-Mental State Examination - MMSE score <18.3)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: CHF was defined as: I) signs (e.g. elevated jugular venous pressure, pulmonary crackles and peripheral edema) and symptoms of HF [New York Heart Association (NYHA) functional class II-IV] in the presence of reduced ejection fraction (LVEF <40%); or II) signs and symptoms of HF (e.g. elevated brain natriuretic peptides and significant structural heart disease/diastolic dysfunction) with mid-range ejection fraction (LVEF 40-49%) or preserved (LVEF ≥50%).
  Patients were diagnosed according to Global initiative for chronic Obstructive Lung Disease (GOLD) criteria (Stage II-IV, C-D); they were in clinically stable condition (no exacerbations in the last 3 months) with optimized stable pharmacological therapy (inhalation therapy with long-acting anticholinergic and/or β2-agonists, inhaled corticosteroids when needed).
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive status | evaluation performed at patient's admission and before discharge (approximately 20 days)
  Addenbrooke's Cognitive Examination III (ACE III) is a 20 minutes screening test, designed for the early detection of cognitive deterioration. It provides a score from 0 to 100 and it analyzes the following five cognitive domains: Attention-Orientation (ACE III-AO = 0-18), Memory (ACE III-M 0 0-26), Verbal Fluency (ACE III-VF = 0-14), Language (ACE III-L = 0-26), and Visuospatial abilities (ACE III-VS = 0-16).
  Frontal Assessment Battery (FAB) is a neuropsychological screening test used to assess executive functions. It is a quick and easy test to administer, its score ranges from 0 to 18, and it is divided into the following six sub-tests: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental dependency.
Changes in Health-related Quality of Life | evaluation performed at patient's admission, before discharge (approximately 20 days) and at 6 months telephone follow-up
  The EQ-5D-5L is a generic quality of life measurement tool. It investigates the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has five levels: 1, no problem; 2, slight problem; 3 moderate problem; 4 severe problem; 5 extreme problem. The second section consists of a Visual Analogue Scale (VAS) from 0 (Worst imaginable health state) to 100 (Best imaginable health state), where the subject is asked to indicate the level of self-perceived wellness.
Changes in psychological characteristics | evaluation performed at patient's admission, before discharge (approximately 20 days) and at 6 months telephone follow-up
  Patient Health Questionnaire-9 (PHQ-9) is a scale used to determine the diagnosis, severity, and subsequent monitoring of depressive illnesses of the patient. It is divided into nine sub-items, to identify depressive symptoms within the last two weeks (following DSM criteria). The final score has a range between 0-27 and it is divided into clinical variability ranges according to a continuum of symptom severity, where scores of 5, 10, 14, and 19 are considered cut-offs for subthreshold, mild major, moderate major, and severe major depression.
  Generalized Anxiety Disorder-7 (GAD) is a questionnaire built to measure the severity of anxiety symptoms in the previous two weeks. The questionnaire consists of 7 items and it organizes the severity of the responses on a 4-point Likert scale. The range scores range from 0 to 21, where scores of 5, 10, and 15 are considered cut-offs for mild, moderate, and severe anxiety, respectively.
Changes in self-reported adherence | evaluation performed at patient's admission, before discharge (approximately 20 days) and at 6 months telephone follow-up
  The Antecedents and Self-efficacy on Adherence Schedule (ASonA) is a self- report schedule aimed to evaluate cognitive, behavioral, and emotional determinants of pharmacological and non-pharmacological adherence. It is a 21-item schedule scored on a 5-point Likert scale (0=not at all, 4=very much). The schedule comprises 3 subscales: Antecedents (ASonA-A), which include health condition and health-related limitations acceptance, social support and knowledge about health condition; Self- efficacy (ASonA-SE), exploring patients' self-care strategies, and patients' ability to adhere to medication assumption and to non-pharmacological recommendations (i.e., physical activity, diet, alcohol consumption, and smoking avoidance); and Affectivity (ASonA-Aff) which measures patients' emotional aspects in relation to the health condition.
Frailty evaluation | evaluation performed at patient's admission
  Frailty Index (FI) is a frailty measurement tool created through a geriatric assessment study including non-institutionalized patients. The variables taken into consideration are mobility, muscle strength, comorbidities, cognitive deficits, mood, anthropometric indices, mini nutritional assessment, and social support. It is made up of 40 items and 17 additional items relating to the Social Support Scale.
Changes in frailty status | evaluation performed at patient's admission, before discharge (approximately 20 days) and at 6 months telephone follow-up
  Clinical Frailty Scale (CFS) is a scale developed in Canada, which is based on clinical judgment only with a score ranging from 1 to 9: 1) Very Fit; 2) Well; 3) Managing Well; 4) Vulnerable; 5) Mildly Frail; 6) Moderately; Frail; 7) Severely frail; 8) Very severely Frail; 9) Terminally Ill [34]. This scale considers clinical data on the subject's cognition, mobility, functional abilities, and comorbidity, which can be collected through the medical history obtained from the patient, the caregiver, and/or other healthcare providers.
Changes in functional performance of the lower extremities | evaluation performed at patient's admission and before discharge (approximately 20 days)
  Short Physical Performance Battery (SPPB) is used to investigate the association between the physical performance and a self-assessed disability by the subjects recruited at a 6-year follow-up. SPPB evaluates the functional capacity of the lower limbs and it consists of three different tests which have been assigned a partial score ranging from 0 to 4.
Changes in mobility | evaluation performed at patient's admission and before discharge (approximately 20 days)
  Timed Up and Go Test (TUG), is a simple test to measure a person's mobility level and requires static and dynamic balancing skills. It measures the time it takes a person to get up from a chair, walk ten feet, turn around, come back to the chair and sit down again.
Changes in functional capacity | evaluation performed at patient's admission and before discharge (approximately 20 days)
  6-minute walking test (6MWT) is a self-limited test used to measure functional exercise abilities in people with HF, Acute Coronary Syndrome, and COPD. It is a test in which the person is asked to walk as fast as possible compatible with his clinical condition for a time of 6 minutes, measuring the meters traveled.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, IRCCS, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vigore M, Granata N, Callegari G, Vaninetti R, Conti S, Maestri R, Piaggi G, Cremonese G, Pierobon A. Frailty and rehabilitation outcome in older patients with cardiorespiratory disease: preliminary multidimensional data. Monaldi Arch Chest Dis. 2022 Dec 1;93(4). doi: 10.4081/monaldi.2022.2447. PMID 36458416
- [Derived] Vigore M, Granata N, Braga SS, Piaggi G, Audifreddi S, Ferrari M, La Rovere MT, Pierobon A. Cognitive impairment, frailty and rehabilitation outcome in older cardiorespiratory patients. DEC_FRAinRIAB: Study protocol. PLoS One. 2022 Aug 4;17(8):e0272132. doi: 10.1371/journal.pone.0272132. eCollection 2022. PMID 35925981